CLINICAL TRIAL: NCT03522883
Title: Acute Effects of Previous Carbohydrate Intake on Perceived Exertion and Muscle Strength in Jiu-jitsu Athletes
Brief Title: Pre-Competition Carbohydrate Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: São Paulo State University (Other)
Collaborators: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Jaqueline Santos Silva, master in physiotherapy, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: SaoPSU_UFMT
Record Dates: First submitted 2018-04-11; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Feeding Behavior
Keywords: Martial Arts
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group control (Placebo Comparator): the subjects will not take any type of nutrient intake
  Interventions: Dietary Supplement: carbohydrate intake prior to exercise
- experimental group 1 (Experimental): carbohydrate intake prior to exercise
  Interventions: Dietary Supplement: carbohydrate intake prior to exercise
- experimental group 2 (Active Comparator): carbohydrate intake prior to exercise
  Interventions: Dietary Supplement: carbohydrate intake prior to exercise

INTERVENTIONS:
Dietary Supplement: carbohydrate intake prior to exercise — Participants will be submitted to carbohydrate supplementation prior to exercise

SUMMARY:
The objective of the present study was to evaluate the MPF and the perception of effort of professional jiu jitsu athletes from carbohydrate intake at different moments. Twelve jiu jitsu athletes participated in the study, being randomly divided into three groups of four participants: Control Group (CG); Experimental group 1 (G1), supplementation immediately before the fight and Experimental group 2 (G2), supplementation 30 minutes before the fight. The FPM measurement was performed with the JAMAR® brand analog hydraulic dynamometer in the pre-fight moments and immediately after the fight. The intensity perception of the effort was verified through the adapted Borg scale after the fight. Regarding the findings on muscle strength, there were different outcomes between the groups analyzed.

DETAILED DESCRIPTION:
The study will be conducted at the "Team Base" training center, located in the western zone of Rio de Janeiro. All procedures were performed under standard conditions (temperature: 21-23 ° C, relative humidity: 40-60%). Participants were previously instructed not to perform vigorous exercise 24 hours prior to data collection and to fast 8 hours prior.

All procedures will be performed in one day. Before the study procedures, participants will be evaluated for anthropometric characteristics using a scale (GAMA ITALY® brand) and a portable stadiometer (Sanny® brand, Personal model). Then, manual palmar grip strength (FPM) will be measured in pre and post fight moments. And, after the fight will also be verified the participants' perception of effort through the adapted Borg scale.

Procedures Fights The struggles (Handori) began respecting the schedules stipulated between the components of the same group. Thus, each fight lasted five minutes, without intervals, where the athletes were instructed to perform dynamic movements, and maintain high movement, aiming to raise the intensity to the maximum during this period.

Carbohydrate Supplementation For the administration of carbohydrate supplementation, the "Advanced Nutrition®" pack containing 30g (1 sachet), energy of 83kcal = 349kJ, carbohydrates 21g, sodium 82mg, vitamin C 4, 2mg and vitamin E 0.90mg.

Palmar Manual Holding Force (FPM) Measurement of the Manual Holding Force (FPM) was performed using the JAMAR® analog hydraulic dynamometer (Asimow Engineering®, USA), with an accuracy of 0.5 kg / f and a maximum capacity of 100 kg / f. Thus, the position suggested by the American Society of Hand Therapists (ASHT) [8] was used, with the participants positioned in a seated position with their hips and knees at 90 ° flexion, shoulder in adduction, elbow flexed at 90 °, wrist and forearm in neutral position. The participant was instructed to perform the greatest possible force and the peak value was subsequently recorded.

Modified Borg Scale Perceived exertion was assessed using the Adapted BORG Scale [7] consisting of an ordinal scale ranging from 0 to 10, where 0 represents none and 10 represents maximum intensity. The following standardized question preceded the application of the scale: "How do you rate the intensity of the exercise performed?" Statistical analysis Mean and standard deviation values were calculated for all variables. The normality of the data was initially analyzed by the Komolgorov-Smirnov procedure. In addition, t-test was used to compare moments and groups. All statistical analysis assumed a significance level of 5%. The analyzes were conducted using the statistical package SPSS (2.0).

ELIGIBILITY:
Inclusion Criteria:

* healthy young people;
* Male, aged 20-45 years, professional jiu jitsu athletes;

Exclusion Criteria:

* musculotendinous lesion or osteoarticular lesion;
* people who take anabolic steroids

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-06-25 (Estimated); Study Completion 2018-08-22 (Estimated)

PRIMARY OUTCOMES:
muscle strength | five minutes
  the muscular force will be measured by means of a manual dynamometer in the dominant upper limb in two moments (pre-fight and post-fight)

SECONDARY OUTCOMES:
Perception of effort | five minutes
  The perception of effort will be measured through a validated scale (BORG), in the moment after competition. It is a graded scale from 0 to 10 that classifies the individual's perception of effort related to the activity performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Ary, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No